CLINICAL TRIAL: NCT05824026
Title: Investigation of the Clinical Performance of Biatain Fiber Ag on Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP357
Record Dates: First submitted 2023-04-11; First posted 2023-04-21 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Partial-thickness Burn
Keywords: infected or risk of infection

STUDY DESIGN:
Intervention Model Description: non-comparative, one-armed, open-labelled, multi-centre study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- main arm (Other): Non comparative - One armed - open labelled Intervention - subjects will wear the test dressing in a two weeks period with planned dressing changes once pr. week.
  Interventions: Device: Gelling fiber wound dressing with silver

INTERVENTIONS:
Device: Gelling fiber wound dressing with silver — intervention involving a wound dressing with silver

SUMMARY:
The goal of this study is to test a new gelling fiber wound dressing with silver on patients with a partial thickness burn wound, which is infected or at risk of infection.

Participants will be asked to wear the test dressing in a two weeks period(+/- 2 days) consisting of 3-4 study visits, and will have the dressing changed once pr. week at the research facility. The wound will be cleaned, assessed and photos will be uploaded to a digital software system.

DETAILED DESCRIPTION:
The clinical investigation is a non-comparative, one-armed, open-labelled, multi-centre study.

The test product, Biatain Fiber Ag is a non-CE-marked gelling fiber wound dressing, containing silver. The product is intended for moist wound healing and exudate management of moderate to high exuding wounds. The product has a classification III, as it contains the active ingredient silver.

The overall purpose of this investigation is to obtain clinical data supporting effectiveness of Biatain Fiber Ag to obtain the CE-mark in EU.

The total study duration for the subject will be approximately two weeks (+/- 2 days), consisting of a two-week test period and 4 study visits (V0/V1, V2 and V3). V3 will also terminate the 2-week study period.

The primary endpoint is percentage of wounds healed within 14 days (≥ 95 % reepithelialisation) The clinical investigation will be conducted in a total of 50 eligible subjects with a partial thickness burn wound that are infected or at risk of infection.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed informed consent
2. Is between 18 -65 years (both included)
3. Is capable of following study procedure (assessed by investigator).
4. Has a partial thickness burn wound
5. Has a burn wound that is infected or at risk of infection (assessed by investigator)
6. The size of burn (including both study wound and non-study injuries) has a Total Body Surface Area (TBSA) less than 10% (assessed by investigator).
7. The wound should fit under a 20x30 cm dressing (600 cm2) or smaller
8. The shape and location of the wound should be suitable for photo capture (assessed by the investigator).
9. Has a wound that has medium to high level of exudate (assessed by the investigator)
10. Is suitable to use the test product for wound treatment (assessed by the investigator).

Exclusion Criteria:

1. Is pregnant/breastfeeding
2. Is currently receiving or has within the past 60 days received radio- and/or chemotherapy (low doses radio- and/or chemotherapy is allowed for other indications than cancer if assessed by investigator not to influence study wound area)
3. Known history of skin sensitivity to any components of the test dressings
4. >72 hours from time of injury
5. Intake of antibiotics within one week before the start of the enrolment
6. Use of chemical debridement
7. Participation in any other clinical studies that can compromise this study treatment (assessed by the investigator).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - North Bristol Southmead Hospital, Westbury, Bristol
  - Buckinghamshire Healthcare NHS Trust, Aylesbury, Buckinghamshire
  - Queen Alexandra Hospital, Portsmouth Hospital University Trust, Cosham
  - Queen Victoria Hospital NHS foundation trust, East Grinstead
  - Newcastle University/The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Arm: Non comparative - One armed - open labelled intervention. Each subject will contribute with one wound (named the study wound), which will be selected at inclusion prior to initiation of treatment.
  Each subject will wear the test dressing in a two weeks period with planned dressing changes once per week.
  The test dressing is a gelling fiber wound dressing with silver applied to the study wounds.
Period: Overall Study
Arm/Group | Main Arm
Started (Safety population/Intention-to-Treat population) | 52
Subjects Where Test Dressing Was Applied at Least Once (Full Analysis Set) | 51
Completed | 43
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: Subjects where test dressing was applied at least once (Full Analysis Set)
Arm/Group | Main Arm
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 49
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 38.9 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 51
Area of subjects' study wound [Mean (Full Range); unit: cm^2] | 52.0 [2 to 177]
Number of Participants with Signs of Infection in the Wound [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Wounds Healed Within 14 Days
Description: The percentage of wounds achieving healing within 14 days (+/- 2 days). A wound was considered healed if re-epithelialization was visually assessed to be 95% or greater.
Time Frame: 2 weeks
Population: Primary analysis was based on the full analysis set for subjects with non-missing data (completers).
  Post hoc sensitivity analysis and supplemental analysis were based on the full analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of wounds healed
Arm/Group | Main Arm
Number analyzed (Participants) | 51
percentage of wounds healed
  Primary analysis (subjects with non-missing data, completers): number analyzed (Participants) | 43
  Primary analysis (subjects with non-missing data, completers) | 83.7 [69.3 to 93.2]
  Post hoc sensitivity analysis (missing data imputed as not healed or using multiple imputation) | 74.8 [60.7 to 85.1]
  Supplemental analysis (missing data imputed as not healed) | 70.6 [56.2 to 82.5]
Statistical Analysis 1: Comparison: Main Arm; Test type: Other; The purpose of the primary analysis was to show non-inferiority to the performance of a historical control (a silver containing gelling fiber) on proportion of wounds healed, 77%, with a non-inferiority margin of 20%. Non-inferiority was demonstrated if the lower limit of the 95% confidence interval is above 57%. An exact confidence interval for the proportion was applied. In the primary analysis missing data was not included. In the post hoc sensitivity analysis missing data was imputed using multiple imputation for 3 wounds where data was assumed to be missing at random, and otherwise imputed as wound not healed. The supplemental analysis addressed a more conservative analysis than performed for the historical control. Hence, no formal non-inferiority criteria was applied for this analysis

ADVERSE EVENTS:
Time Frame: 2 weeks (+/- 2 days)
Arm/Group | Main Arm
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 1/52
Other Adverse Events (participants affected / at risk) | 10/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Arm (N=52)
Rash (Immune system disorders) | 1 (1) — Not related to investigational device
Hypotension (Cardiac disorders) | 1 (1) — Not related to investigational device
Swollen feet and ankles (Vascular disorders) | 1 (1) — Not related to investigational device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Arm (N=52)
Severe pain from dressed burn wound (Skin and subcutaneous tissue disorders) | 1 (1) — Possibly related to investigational device
Dressing difficult to remove/wound bleeding after dressing removal (Skin and subcutaneous tissue disorders) | 5 (5) — Related to investigational device
Pain at the site where dressing had been applied (Skin and subcutaneous tissue disorders) | 1 (1) — Related to investigational device
Wound infection (not study wound) (Infections and infestations) | 2 (2) — Not related to investigational device
Chest infection (Infections and infestations) | 1 (1) — Not related to investigational device
Diarrhoea (Gastrointestinal disorders) | 1 (1) — Not related to investigational device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT05824026/Prot_SAP_000.pdf